CLINICAL TRIAL: NCT04575285
Title: Using EEG to Predict Depression Treatment Response to Repetitive Transcranial Magnetic Stimulation (rTMS) in Patients With Major Depression
Brief Title: Using EEG to Predict Depression Treatment Response to rTMS in Patients With Major Depression
Status: Withdrawn | Type: Observational
Why Stopped: Study was closed due to lack of resources
Sponsor: Baptist Health South Florida (Other)
Collaborators: Florida International University (Other)
Responsible Party: Sponsor
Other Study IDs: TMS Depression
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2022-03

CONDITIONS: Major Depression; Repetitive Transcranial Magnetic Stimulation
Keywords: rTMS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Electroencephalogram (EEG): All participants will undergo EEG recording at baseline and end of treatment for a duration of 10-20 minutes per session.
  Interventions: Diagnostic Test: Electroencephalogram (EEG)

INTERVENTIONS:
Diagnostic Test: Electroencephalogram (EEG) — EEG measures brain activity by recording the spontaneous brain electrical activity and evoked responses non-invasively from the scalp. Reusable Tangle Free 10mm EEG Cup Electrodes will be placed on the subject's scalp using the 10-20 system montage.

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a promising, novel, non-invasive therapy for depression. The study is looking at changes in specific electroencephalogram parameters in depressed patients treated with rTMS can serve as predictors of depression treatment response among cancer patents undergoing rTMS treatment of depression.

DETAILED DESCRIPTION:
The study will be a prospective, single arm trial in which a set of patients who will be treated for major depression using Repetitive Transcranial Magnetic Stimulation (according to FDA approved rTMS standard care practices) also will undergo EEG recording before Repetitive Transcranial Magnetic Stimulation treatment begins, and at the completion of treatment. The Hamilton Depression Rating Scale will be given to participants by the neuropsychiatrist at baseline and weekly intervals till the completion of treatment.

The neuropsychiatrist investigators expect to see about 12 patients per year who meet treatment criteria for Repetitive Transcranial Magnetic Stimulation. Therefore, it is expected to recruit 24 subjects into the research study over a two-year period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer
* Comorbid diagnosis of major depressive disorder
* Age ≥ 18 years
* Baseline Hamilton Depression Rating Scale (HDRS) score ≥ 18
* Failed one or more adequate antidepressant trials (including selective serotonin reuptake inhibitors or SSRIs, selective norepinephrine reuptake inhibitors or SNRIs, tricyclic antidepressants or TCAs). A failed treatment response may be due to lack of antidepressant efficacy or intolerable side effects.

Exclusion Criteria:

* History of seizure or epilepsy
* History of concussion
* History of bipolar disorder
* Comorbid psychotic disorder
* Primary brain tumor or metastasis to brain
* Active comorbid substance use disorder
* History or current diagnosis of dementia
* Current pregnancy
* Unable to attend regular treatment sessions
* Any other condition in which a physician investigator feels may subject the participant to undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be treated for major depression using rTMS (according to standard care)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale score | baseline, and weekly until study completion, which can be up to 6 weeks
  Hamilton Depression Rating Scale is used to measure severity of depression on a scale from 0 (no depression) to 52 (most severe depression).

SECONDARY OUTCOMES:
Electroencephalograph (EEG) scalp signal changes over time | baseline, end of treatment, which can be up to 6 weeks
  Change in brain activity as measured by the EEG in microvolts.Scalp EEG signals will be processed in order to compare EEG brain connectivity and Frontal alpha asymmetry index (FAA).

CONTACTS AND LOCATIONS:
Overall Officials: Geetha Nampiaparampil, MD, Principal Investigator — Miami Cancer Institute (MCI) at Baptist Health, Inc.
Locations (1):
- Starlie C Belnap, Miami, Florida, United States

REFERENCES:
- See also: Miami Neuroscience Institute — https://neuroscience.baptisthealth.net/miami-neuroscience-institute